CLINICAL TRIAL: NCT03139747
Title: UPCC 36315 A Phase II Study Of Everolimus (RAD001) And Lenvatinib (E7080) In Patients With Metastatic Differentiated Thyroid Cancer Who Have Progressed on Lenvatinib Alone
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual reevaluating feasibility
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 36315
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — lenvatinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Lenvatinib; Drug: Everolimus

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib is an anti-cancer drug for the treatment of certain kinds of thyroid cancer, and potentially for other cancers as well. It was developed by Eisai Co. and acts as a multiple kinase inhibitor against the VEGFR1, VEGFR2 and VEGFR3 kinases.
Drug: Everolimus — It is currently used as an immunosuppressant to prevent rejection of organ transplants and in the treatment of renal cell cancer and other tumours. Much research has also been conducted on everolimus and other mTOR inhibitors as targeted therapy for use in a number of cancers.

SUMMARY:
This is a Phase 2 Study of Everolimus and Lenvatinib in patients with metastatic differentiated thyroid cancer who have progressed on lenvatinib alone. Patient will have imaging, lab test and physical exams

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years old or older.
* ECOG performance status < 2 (Appendix 1).
* Patients must have histologically confirmed differentiated thyroid cancer, that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Patients may have received multiple treatments of radioactive iodine. Patients may have received one or more prior MKI treatments that are not lenvatinib (note: all patients will have been required to have had lenvatinib for entry, see below). At least 4 weeks must have elapsed since prior non-lenvatinib MKI treatment.
* Patients are eligible immediately following progression on lenvatinib. Patients must have had documented progression while on the prior treatment with lenvatinib and must have had a minimum of stable disease for 4 months.
* Measurable disease defined as at least one malignant lesion that can be accurately and serially measured in at least one dimension (longest diameter to be recorded) using conventional methods (CT, MRI, x-ray, PE) (diameter > 20 mm) or spiral CT (diameter > 10 mm).
* Life expectancy greater than 3 months.
* Adequate organ function that has been determined within 14 days prior to enrollment, defined as:
* Leukocyte count > 3,000/uL; Absolute neutrophil count (ANC) > 1,500/mm3, platelets > 75,000/mm3, and hemoglobin > 9 g/dl.
* Serum creatinine < 1.5 times ULN, or 24-hour creatinine clearance > 75 cc/min. (Note: creatinine clearance need not be determined if the baseline serum creatinine is within normal limits).
* Serum bilirubin < 2.0mg/dL; ALT and AST < 2.5 ULN;
* INR < 2.0 or a PT/PTT within normal limits. Exception allowed for patients receiving anti-coagulation treatment with an agent such as warfarin or heparin who may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of lenvatinib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Intellectual, emotional, and physical ability to comply with oral medication.
* Ability to understand and the willingness to sign a written informed consent
* Signed informed consent obtained prior to any screening procedures.

Exclusion Criteria:

* Patients who have had any intervening systemic cancer treatment since the prior lenvatinib treatment.
* Patients with significant medical disease including: uncontrolled congestive heart failure; active symptoms of coronary artery disease, uncontrolled seizure disorder; active infection; uncontrolled diabetes mellitus; requirement for chronic high dose corticosteroid treatment (Topical or inhaled corticosteroids are allowed); requirement for concurrent immunosuppressive drug(s); active autoimmune disease.
* Patients with organ allografts.
* Patients with uncontrolled BP prior to the start of treatment
* Patients with known HIV-infection (HIV testing is not required for participation).
* Pregnant or nursing (lactating) women;
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after. Highly effective contraception methods include any of the following:
* Use of oral, injected or implanted hormonal methods of contraception or;
* Placement of an intrauterine device (IUD) or intrauterine system (IUS);
* Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
* Total abstinence or;
* Male/female sterilization. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential. Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients with a history of second cancer (except adequately non-melanoma skin cancer, in situ treated cancer of the cervix, uterus, colon cancer or melanoma, any benign cancer for which the patient does not require treatment, or any other cancer for which the patient has been disease-free for three or more years).
* Patients who have received live attenuated vaccines within 1 week of start of Everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines;
* Patients with uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
* Patients with known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus);
* Patients who have any severe and/or uncontrolled medical conditions such as:
* unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to start of Everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
* Symptomatic congestive heart failure of New York heart Association Class III or IV
* active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA),
* known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air),
* active, bleeding diathesis;
* Patients requiring chronic treatment with corticosteroids or other immunosuppressive agents. Topical or Topical or inhaled corticosteroids are allowed;
* Patients with a known history of HIV seropositivity;
* Use of any experimental therapy within 4 weeks prior to baseline evaluations done prior to enrollment (with the exception of lenvatinib which may be continued until treatment start). Therefore, all experimental treatments other than lenvatinib must be discontinued 4 weeks prior to baseline studies or enrollment.
* Patients with known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption;
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study;
* Patients already scheduled to have a lymph node dissection may have the procedure performed on-study as long as the lymph nodes are not followed as part of RECIST criteria and all study medications are held from three days prior to the procedure to one week following or until deemed safe by the treating physician
* Patients with carcinomatous meningitis are excluded from the study. Patients with treated sites of leptomeningeal disease may be included at the discretion of the principal investigator.
* Patients who are not expected to tolerate a starting dose of 18mg lenvatinib and 5mg everolimus daily will not be considered eligible for the study.
* Excludedtherapies and medications, previous or concomitant:
* Anticancer chemotherapy or immunotherapy during the study or within 4 weeks prior to the first dose of the study drug with the exception of lenvatinib
* Radiotherapy for the treatment of a symptomatic (e.g. bone metastasis) as clinically indicated is allowed as long as it is not evidence of progressive disease and is not required to be measured as a target lesion per RECIST Biological response modifiers, such as G-CSF, within 3 week prior to study entry. (G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator; however they may not be substituted for a required dose reduction).
* Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study.
* Investigational drug therapy outside of this trial during or within 4 weeks prior the screening assessment.
* Use of ketoconazole, itraconazole, and ritonavir.
* Use of carbamazepine, phenytoin, phenobarbital.
* Use of grapefruit juice products.
* Use of cyclosporin.
* Use of coumadin is discouraged, and patients where possible should be switched to lovanox.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with progression free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Brose, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States